CLINICAL TRIAL: NCT05092971
Title: Identifying Decision Making Parameters in Healthy Volunteers (HV) and Anxiety Patients (AD)
Brief Title: Identifying Decision Making Parameters in Healthy Volunteers and Anxiety Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10000378; 000378-M
Record Dates: First submitted 2021-10-23; First posted 2021-10-26 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2022-07-28

CONDITIONS: Anxiety; Healthy Volunteers
Keywords: functional magnetic resonance imaging (fMRI); multi-arm bandit task; anxiety volunteers; Healthy Volunteers
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Anxiety patient (Experimental): Participants with anxiety completed computer tasks. They were given different choices and had to make choice(s). The objective was to find the optimal choice by sampling through the choices. They received an unpleasant or pleasant stimulus based on their choice(s). They repeated these tasks many times.
  Interventions: Device: Shock or startle device
- Healthy volunteer (Experimental): Healthy volunteers completed computer tasks. They were given different choices and had to make choice(s). The objective was to find the optimal choice by sampling through the choices. They received an unpleasant or pleasant stimulus based on their choice(s). They repeated these tasks many times.
  Interventions: Device: Shock or startle device

INTERVENTIONS:
Device: Shock or startle device — Shock and startle devices were used as aversive stimulus (shock and startle)

SUMMARY:
Background:

Research has shown that anxiety affects more than feelings. It also affects behavior. Researchers want to learn how the brain and body respond to unexpected threats. They want to see if probable pleasant or unpleasant events change decisions.

Objective:

To better understand how changes in anxiety are associated with changes in decision-making.

Eligibility:

Adults aged 18-50 with generalized anxiety disorder, seasonal affective disorder, or panic disorder. Healthy volunteers are also needed.

Design:

Participants will be screened under protocol #01-M-0254.

Participants will complete surveys about their anxiety, risk-taking, and curiosity.

Participants will complete a computer task. They will be given different choices. They will make a choice. They will receive an unpleasant or pleasant stimulus based on their choice. They will repeat this task many times.

Most participants will do the task in the clinic. The unpleasant stimulus will be electric shock and acoustic startle. They will receive electric shocks through electrodes placed on their arm or fingers. They may hear loud noises through headphones. Their eyeblinks will be recorded with electrodes placed under their eye. Their heart rate and skin conductance activity will be collected with electrodes as well.

Some healthy volunteers will do the task during a functional magnetic resonance imaging scan. They will lie on a table that slides in and out of a scanner. A coil will be placed over their head. The unpleasant stimulus will be electric shock, given as stated above. The scanner will record their brain activity. Their breathing and pulse rate will be recorded as well.

Participation will last for 3-4 hours.

DETAILED DESCRIPTION:
Study Description:

This study s goal is to identify parameters of interest in decision making in the context of anxiety disorders, using theoretical models in healthy volunteers (HV) and anxiety patients (AD). Participants are asked to complete a decision-making task, namely the Multi-armed Bandit Task.

The study will be conducted in the clinic. Participants (HV and AD) are asked to fill out questionnaires and complete the Multi-armed Bandit Task. An electric shock is used as the aversive stimulus. Monetary reward is used as the reward stimulus. Additionally, physiological signals (Heart rate, skin conductance activity, startle) are collected during the course of the task. In addition, in a pilot study, participants startle responses for varying shock parameters are recorded and analyzed.

Objectives:

The primary objective of this study is to use theoretical models in healthy volunteers (HV) and patients with an anxiety disorder (AD) to better understand how changes in anxiety are associated with changes in decision making. In addition, this study will ascertain whether decision making parameters correlate with certain behavioral measures such as trait and state anxiety using (i) questionnaires, (ii) physiological measures.

Endpoints:

The primary endpoint of this study is a significant difference in model derived parameters between experimental manipulations (conditions) and/or population groups. The parameters of interest include: 1) Learning Rate, 2) Exploration parameter, 3) Discount rate, 4) Loss aversion, 5) Inverse Temperature.

The secondary endpoints are a significant correlation between functions of model derived parameters and behavioral and/or physiological measures of anxiety including:

1. Questionnaire scores
2. Startle
3. Skin conductance

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Male or female, aged 18-50, inclusive
3. Patients only: Primary Diagnostic and Statistical Manual (DSM) 5 diagnoses of an anxiety disorder (GAD, social anxiety disorder (SAD), panic disorder)

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Non-English speaking individual
2. Pregnancy or positive pregnancy test
3. Any significant medical or neurological problems as determined by investigators (e.g.cardiovascular illness, respiratory illness, neurological illness, seizure, etc.)
4. Current or past serious mental disorders (e.g., bipolar or psychotic disorders) (except for anxiety and depressive disorders in patients)
5. Current alcohol or substance use disorder
6. History of moderate or severe alcohol or substance use disorder within one year prior to screening
7. Current or past significant organic central nervous system disorders as determined by investigators, including but not limited to seizure disorder or neurological symptoms of the wrist and arm (e.g., carpal tunnel syndrome) for shocks to be delivered on affected arm.
8. Positive urine toxicology screen at screening visit under 01-M-0254
9. Employees of National Institute of Mental Health (NIMH) or an immediate family member of a NIMH employee.
10. Healthy volunteers only: Current DSM-5 disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maryland Pao, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will be shared to a repository. Identified individual participant data will not be shared.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000378-M.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anxiety Patient | Healthy Volunteer
Started | 20 | 31
Completed | 20 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anxiety Patient | Healthy Volunteer | Total
Number analyzed (Participants) | 20 | 31 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 31 | 51
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 1 | 13 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 15 | 30 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 8 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 12 | 17 | 29
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Difference in Learning Rate
Description: Learning rate is a hyperparameter that quantifies the degree to which subjects update their beliefs in response to feedback. The outcome examined the difference in learning rate between experimental manipulation (condition) and population (healthy and anxiety subjects). During the multi-arm bandit task, participants choose from a set of choices and update their belief of the value of the choices based on prior choices with some choices having a higher probability of shock (punishment) than reward.
  The changes in learning rate were measured using the learning rate algorithm. The difference in learning rate was analyzed using a 2-way ANOVA with condition and population.
  The learning rate (α) range between 0 and 1. The higher the value, the faster rate of learning. However, a higher learning rate may also result in lower generalization capability.
Time Frame: End of experiment (3-4 hours in a single day visit)
Population: Analysis included all participants who completed the study.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Anxiety Patient | Healthy Volunteer
Number analyzed (Participants) | 20 | 31
unitless | 0.009 (0.0315) | 0.0058 (0.037)

ADVERSE EVENTS:
Time Frame: One day
Arm/Group | Anxiety Patient | Healthy Volunteer
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/31
Other Adverse Events (participants affected / at risk) | 0/20 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT05092971/Prot_SAP_000.pdf